CLINICAL TRIAL: NCT01904578
Title: The Effect of Acupressure on Sleep Quality in Menopausal Women
Brief Title: The Efficacy of Acupressure on Sleep Quality in Menopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Abedian, Instructor of Midwifery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: treatment
Record Dates: First submitted 2012-07-07; First posted 2013-07-22 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2010-02

CONDITIONS: Poor Quality Sleep
Keywords: Menopause; Sleep quality; Acupressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- true acupressure (Experimental): Massage the effective pressure points as a self-care method at home [ Four acupoints were chosen for subjects in the acupressure group. They were Shenmen on the wrist crease, Sanyinjiao point (SP6) on both feet, Fengchi on the hairline of the back neck (occipital area)and Yintang, at the top of the nose on the centre line between the ends of the eyebrows] for 10 minutes. It was done 1 to 2 hours before sleeping, each night (except Fridays) by circular massage with a 1 Cm circle diameter.
  Interventions: Other: true accupressure
- sham acupressure (Sham Comparator): Massage the sham pressure points as a self-care method at home for 10 minutes. It was done 1 to 2 hours before sleeping, each night (except Fridays) by circular massage with a 1 Cm circle diameter.
  Interventions: Other: sham acupressure
- control (No Intervention): The control group only received the weekly control of blood pressure and speech communication .

INTERVENTIONS:
Other: true accupressure — Four acupoints were chosen for subjects in the acupressure group. They were Shenmen on the wrist crease, Sanyinjiao point (SP6) on both feet, Fengchi on the hairline of the back neck (occipital area)and Yintang, at the top of the nose on the center line between the ends of the eyebrows.
  Arms: true acupressure
Other: sham acupressure — Non-acupoints, which were 1 to 3 traditional Chinese unit of length (CUN) away from true acupoints, were used in sham acupressure group.These points were out of the route of energy
  Arms: sham acupressure

SUMMARY:
Sleep disorder is a common problem in menopausal women and the decrease in the sleep leads to poor daily activity. Traditional Chinese acupressure is a noninvasive, effective and safe technique that can be easily taught to menopausal women so that they apply it as a self-care method and a manager of sleep disruption. The purpose of the present study was to evaluate the effectiveness of acupressure on sleep quality of postmenopausal women.This double blind randomized clinical trial was performed on 120 qualified menopausal women at the age of 41-65 years; and sleep quality was measured with Pittsburgh Sleep Quality Index (PSQI ).Participants were randomly assigned to an acupressure group, a sham acupressure group and a control group by two time randomized method (systematic and simple randomized). These interventions were carried out for 4 consecutive weeks. Participants in acupressure group and sham acupressure group learned to carry out acupressure technique as a self care at home with the simultaneous massage techniques that were to be performed 2 hours before sleep, whereas only conversation was used in the control group. The statistical software package for social science (SPSS) Version 17 was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* spending at least 12 months after amenorrhea or follicle stimulating hormone
* (FSH) Serum level ≥ 40,
* healthy of the pressure points,
* having a full consciousness
* having an acceptable ability of listening
* speaking to receive training
* doing the self- care techniques at home,
* no mental and physical disorders,
* getting a score higher than 5 from the Pittsburgh Sleep Quality Index (PSQI)
* able to sit for about 30 minutes.

Exclusion Criteria:

* having specific eating diets,
* addicted to narcotic drugs,
* using the drugs causing sleep disorders,
* suffering from special disease,
* taking hormonal drugs during 3 last months,
* using herbal medicine to improve the menopausal symptoms,
* BMI higher than 30,
* having the moderate and severe depression based on Beck Depression Inventory,
* feeling of severe tiredness/ fatigue and anxiety,
* having circular job specially night job
* lack of cooperation with researchers.

Ages: 41 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
treatment of quality of sleep | 4 consecutive weeks
  treatment of quality of sleep by acupressure.sleep quality was measured with Pittsburgh Sleep Quality Index (PSQI ).